CLINICAL TRIAL: NCT07053904
Title: A Phase I, Open-Label Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Sequential Treatment With P1101 and P1801 in Patients With Advanced Solid Tumors
Brief Title: Phase I Open-Label Study of P1101 Followed by P1801 in Advanced Solid Tumors
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaEssentia (Industry)
Collaborators: Efficient Pharma Management Corp. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C23-101
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort 1: Sequential 6 doses of P1101 followed by P1801 (0.3 mg/kg, Q2W) (Experimental): Sequential 6 doses of P1101 450 mcg, Q2W; followed by P1801 0.3 mg/kg, Q2W
  Interventions: Drug: Sequential use of P1101 and P1801
- Cohort 2: Sequential 6 doses of P1101 followed by P1801 (0.75 mg/kg, Q2W) (Experimental): Sequential 6 doses of P1101 450 mcg, Q2W; followed by P1801 0.75 mg/kg, Q2W
  Interventions: Drug: Sequential use of P1101 and P1801
- Cohort 3: Sequential 6 doses of P1101 followed by P1801 (1.5 mg/kg, Q2W) (Experimental): Sequential 6 doses of P1101 450 mcg, Q2W; followed by P1801 1.5 mg/kg, Q2W
  Interventions: Drug: Sequential use of P1101 and P1801
- Cohort 4: Sequential 6 doses of P1101 followed by P1801 (2.0 mg/kg, Q2W) (Experimental): Sequential 6 doses of P1101 450 mcg, Q2W; followed by P1801 2.0 mg/kg, Q2W
  Interventions: Drug: Sequential use of P1101 and P1801
- Cohort 5: Sequential 6 doses of P1101 followed by P1801 (3.0 mg/kg, Q2W) (Experimental): Sequential 6 doses of P1101 450 mcg, Q2W; followed by P1801 3.0 mg/kg, Q2W
  Interventions: Drug: Sequential use of P1101 and P1801

INTERVENTIONS:
Drug: Sequential use of P1101 and P1801 — Sequential use of ropeginterferon alfa-2b and P1801 (anti PD-1 antibody drug)

SUMMARY:
The goal of this clinical trial is to learn the safety of sequential treatment with P1101 and P1801 in advanced solid tumors. It will also learn the maximum tolerated dose (MTD) of P1801. The main questions it aims to answer are:

To evaluate the safety and tolerability of sequential treatment with P1101 and P1801 in patients with advanced solid tumors.

To determine the maximum tolerated dose (MTD) of P1801.

Participants will:

Ttreated by 6 doses of P1101 once per 2 weeks (Q2W) at 450 mcg and then followed by the treatment with P1801 Q2W at the pre-determined dose level by cohort during each 28-day treatment cycle in the Dose Escalation Phase (Cohort 1-5).

Once the MTD have been declared and for further characterize safety and clinical activity, additional patients with RCC or CRC will be enrolled into the tumor-specific expansion cohorts to receive the sequential administration of 6 doses of P1101 Q2W at 450 ug followed by P1801 Q2W at MTD.

Patients will visit the clinic every two weeks during the treatment period for drug administration and physical examinations.

All patients must complete the safety follow-up visits at the 30-, 90-, and 150-day after the last dose of study treatment.

Upon completion of the safety follow up, patients will be followed for survival every 12 weeks until death or until the end of the study is reached, unless they withdraw consent or are lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to provide written informed consent;
2. Age ≥18 years;
3. Patients with histologically or cytologically confirmed metastatic or locally advanced solid tumors who have progressed despite standard therapy or are intolerant to standard therapy or for whom there is no standard therapy;
4. Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 1 at trial entry and an estimated life expectancy of at least 3 months;
5. Dose Escalation Phase: Patients with an advanced solid tumor, including, but not limited to RCC and CRC; Dose Expansion Phase: Patients with RCC or CRC;
6. Prior chemotherapy or immunotherapy must have been completed at least 4 weeks before screening, and all adverse events have either returned to baseline or stabilized;
7. Prior systemic radiation therapy must have been completed at least 4 weeks before screening;
8. Normal fundoscopic examination by ophthalmologist at screening; major fundoscopic findings including, but not limited to retinal exudates, hemorrhage, detachment, neovascularization, papilloedema, optic atrophy, microaneurysms and macular changes;
9. Patient who has normal laboratory values relevant to thyroid function.

Exclusion Criteria:

1. Concomitant disease or condition that could interfere with the conduct of the study in the opinion of the Investigator;
2. Patients requiring chronic treatment with systemic corticosteroids in excess of 10 mg daily of prednisone or equivalent or receiving any systemic immunosuppressive medication will be excluded; while topical, inhaled, nasal and ophthalmic steroids are not prohibited;
3. Patients with an active autoimmune disease, a documented history of autoimmune disease or syndrome or asthma that requires systemic steroids or immunosuppressive agents;
4. Untreated or symptomatic brain metastasis;
5. Subjects with any of the following laboratory test or complications:

   * Creatinine > l.5 X Upper Limit of Normal (ULN);
   * Absolute neutrophil count (ANC) < 1,500/μL;
   * Platelet count < 100,000/μL;
   * Hemoglobin < 9 g/dL;
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 X ULN (> 5 X ULN if liver metastasis), or total bilirubin > 1.5 X ULN
   * international normalized ratio (INR) or activated partial thromboplastin time (aPTT) > 1.5 X ULN;
   * uncontrolled diabetes mellitus (HbA1c ≥7.4%);
6. Any presence of poorly controlled major psychiatric (including but not limited to those with severe depression, severe bipolar disorder, schizophrenia, suicidal ideation or history of suicidal attempt);
7. Any presence of poorly controlled cardiovascular (including but not limited to those with uncontrolled hypertension, New York Heart Association (NYHA) class 2 congestive heart failure, uncontrolled arrhythmia, severe coronary arterial stenosis, unstable angina); or with history of stroke or acute myocardial infarction within 3 years prior to screening;
8. Female subjects or the spouse of male subjects, with child-bearing potential who are unwilling or unable to practice any highly effective methods of contraception, defined as vasectomy in men, tubal ligation in women, or use of condoms and spermicides, or birth control pills, or intrauterine devices from 28 days prior to Day 1 until the final follow up visit;
9. Patients who are pregnant, who have a possibility of being pregnant or who desire to become pregnant during the study period;
10. Lactating women;
11. History of hypersensitivity reactions to the active ingredients or any excipient of the study drugs; or history of severe hypersensitivity reactions to other monoclonal antibodies;
12. Use investigational drug of other clinical trials within 4 weeks prior to screening;
13. History of drug-induced pneumonitis or current pneumonitis;
14. Active infection requiring systemic antibiotic therapy;
15. Patients with HBV DNA ≧ 2,000, positive HCV RNA, or known human immunodeficiency virus (HIV) infection;
16. Patients with Common terminology criteria for adverse events (CTCAE) Grade ≥ 3 cardiac disease or with a history of cardiac arrest;
17. Receive any vaccination within 4 weeks prior to screening;
18. Use telbivudine within 4 weeks prior to screening or those will use telbivudine after screening;
19. Use of prohibited medication or herbal remedies within 4 weeks prior to screening;
20. History of CTCAE Grade ≥3 immune-related adverse event (AE) that was considered related to prior immune-modulatory therapy or any immune-related AEs that required immunosuppressive therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicities (DLTs) | P1801 treatment cycle is comprised of 2 doses of P1801 administered on Day 1 (CnD1) and Day 15 (CnD15) at each cycle. Eligible patients will be monitored for the occurrence of DLTs during a 28-day period (Cycle 1) after the first administration of P1801.
  Incidence of Dose-Limiting Toxicities (DLTs) of P1801
MTD of P1801 | highest dose level at which no more than 1 out of 6 patients experiences a DLT during the 28-day observation period.
  The MTD is defined as the highest dose level at which no more than 1 out of 6 patients experiences a DLT during the 28-day observation period.

CONTACTS AND LOCATIONS:
Locations (2):
- Taiwan (2):
  - Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, New Taipei City
  - Taipei Medical University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No